CLINICAL TRIAL: NCT02621554
Title: Impact of Resveratrol on Brain Function and Structure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Planck Institute for Human Cognitive and Brain Sciences (Other)
Collaborators: University of Leipzig (Other); Evolva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: resveratrol_mpi_01
Record Dates: First submitted 2015-11-06; First posted 2015-12-03 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Memory; Resveratrol; elderly; cognition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resveratrol supplementation (Experimental): Dietary Supplement: Resveratrol
  Interventions: Dietary Supplement: resveratrol supplementation
- placebo supplementation (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: resveratrol supplementation — 6 months of resveratrol supplementation
  Arms: resveratrol supplementation
Dietary Supplement: Placebo — 6 months of placebo intake
  Arms: placebo supplementation

SUMMARY:
The study will investigate whether resveratrol could provide positive effects on memory and brain structures and functions in healthy elderly participants.

DETAILED DESCRIPTION:
Cell and animal studies postulated various beneficial effects of resveratrol, ranging from a reduction of inflammatory processes and the treatment of cancer to the prevention of cardiovascular diseases and stroke. With regard to cognitive decline, rodent models for Alzheimer's disease (AD) showed improved learning and decelerated hippocampal neurodegeneration after intake of resveratrol.

Animal and first human studies provided evidence that resveratrol might serve as an easy, cost-effective option to develop novel prevention and treatment strategies against age-associated cognitive decline. To test this hypothesis, the researchers study general brain structure and function on healthy older individuals (> 60years old).

ELIGIBILITY:
Inclusion Criteria:

* subjects who are healthy or with subjective memory complaints
* older than 60 years old
* normal to overweight participants (BMI: 22-40 kg/sqm)

Exclusion Criteria:

* dementia
* Psychiatric diseases
* severe untreated internal diseases
* diabetes
* younger than 60 years
* BMI < 22 or >40

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Verbal Learning Task Scores at 6 months | Baseline (timepoint 0), after 6 months (timepoint 6 months)

SECONDARY OUTCOMES:
Change from baseline Verbal Learning Task Scores at 12 months | after 12 months (timepoint 12 months)
Mini Mental State Examination | Baseline (timepoint 0), after 6 months (timepoint 6 months) and after 12 months (timepoint 12 months)
Structural changes on the brain MRI images | Baseline (timepoint 0), after 6 months (timepoint 6 months) and after 12 months (timepoint 12 months)
Functional changes on the brain MRI images | Baseline (timepoint 0), after 6 months (timepoint 6 months) and after 12 months (timepoint 12 months)
Plasma biomarkers | Baseline (timepoint 0), after 6 months (timepoint 6 months) and after 12 months (timepoint 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Arno Villringer, Prof., Study Chair — Max Planck Institute for Human Cognitive and Brain Sciences; Arno Villringer, Study Director — Max Planck Institute for Human Cognitive and Brain Sciences; Veronica Witte, Study Director — Max Planck Institute for Human Cognitive and Brain Sciences; Veronica Witte, Principal Investigator — Max Planck Institute for Human Cognitive and Brain Sciences
Locations (1):
- Department of Neurology, Max Planck Institute for Human Cognitive and Brain Sciences, Leipzig, Germany

REFERENCES:
- [Derived] Huhn S, Beyer F, Zhang R, Lampe L, Grothe J, Kratzsch J, Willenberg A, Breitfeld J, Kovacs P, Stumvoll M, Trampel R, Bazin PL, Villringer A, Witte AV. Effects of resveratrol on memory performance, hippocampus connectivity and microstructure in older adults - A randomized controlled trial. Neuroimage. 2018 Jul 1;174:177-190. doi: 10.1016/j.neuroimage.2018.03.023. Epub 2018 Mar 13. PMID 29548848
- Available data/document: Statistical Analysis Plan — https://drive.google.com/open?id=0Bx6LS4H2DroFNnVaQWlTakh5dEU
- Available data/document: Statistical Analysis Plan — https://drive.google.com/open?id=0Bx6LS4H2DroFazRhT1hZVm41RzA — 05.01.2017 updated because of an amendment of ethnic proposal.